CLINICAL TRIAL: NCT01525498
Title: Urinary Bladder Catheterization Following Sacrocolpopexy
Brief Title: Foley Catheterization Following Sacrocolpopexy
Status: Withdrawn | Type: Observational
Why Stopped: No subject accrual
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Other Study IDs: Foley
Record Dates: First submitted 2012-01-19; First posted 2012-02-03 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Pelvic Organ Prolapse; Catheter Infection; Urinary Retention
Keywords: Pelvic Organ Prolapse; Catheterization; Urinary tract infection; Urinary retention
MeSH Terms: conditions — Pelvic Organ Prolapse; Urinary Retention; Urinary Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1 day catheter removal: Participants randomized to group 1 will have their catheter removed 1 day after surgery.
- 2 day catheter removal: Participants randomized to group 2 will have their catheter removed 2 days after surgery.

SUMMARY:
The objective of this study is to prospectively evaluate the effects of early versus delayed removal of transuretheral catheters following sacrocolpopexy. The investigators specific aim is to determine the optimal time of removal of an indwelling transurethral catheter postoperatively in an effort to reduce the risk of postoperative urinary retention and urinary tract infection associated with catheter use. The investigators hypotheses are as follows:

Hypothesis 1: Longer duration of postoperative catheter use will result in decreased postoperative urinary retention.

Hypothesis 2: Shorter duration of postoperative catheter use will result in lower incidence of urinary tract infection.

DETAILED DESCRIPTION:
Patients scheduled to undergo sacrocolpopexy for pelvic organ prolapse at the University of Oklahoma Health Sciences Center will be recruited for this study. Written informed consent will be obtained from all participants prior to the scheduled surgery and before the randomization process. This study will contain two arms, each with two groups. The first arm will have participants receiving sacrocolpopexy for pelvic organ prolapse; the second arm will consist of participants receiving sacrocolpopexy plus a concomitant procedure for stress urinary incontinence. Each participant will be assigned to the arm that matches their scheduled procedure; they will then be randomized into one of the two study groups within that arm. Randomization will be performed by placing note cards in sealed envelopes with "Group A" or "Group B" listed on the card. One envelope will be placed with each participant's preoperative packet and opened on the day of surgery after the operation is complete.On the date of the procedure, a urinalysis will be performed prior to the routine administration of prophylactic antibiotics. At the beginning of the procedure, a transurethral catheter will be placed as is routine for this procedure. At the conclusion of the procedure, the sealed envelope containing the participant's group designation will be opened and she will be assigned to one of two groups. Group A participants will have their catheter removed on postoperative day 1 and Group B will have their catheter removed on postoperative day 2.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 21
* Scheduled to undergo sacrocolpopexy at the University of Oklahoma Health Sciences Center

Exclusion Criteria:

* Age < 21
* Elevated postvoid residual measurement on preoperative exam
* History of urinary retention
* Medical or surgical indication for prolonged catheterization
* History of neurologic problems

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The projected sample size is 584 participants. Participants will be drawn from the University of Oklahoma Urogynecology clinics. Our catchment area includes OU Physicians clinic (private clinic) and Presbyterian Professional Building (resident clinic).
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-08; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Urinary retention following catheter removal | 2 days
need for repeat catheterization | 2 days
Presence of bacteriuria at catheter removal | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Abbas Shobeiri, MD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States